CLINICAL TRIAL: NCT02952001
Title: MAGNOLIA: Multi-Center, Non-Interventional Extension Study of the Safety and Efficacy of CLS-TA for the Treatment of Macular Edema Associated With Non-Infectious Uveitis
Brief Title: MAGNOLIA: Extension Study of Patients With Non-infectious Uveitis Who Participated in CLS1001-301
Status: Completed | Type: Observational
Sponsor: Clearside Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLS1001-303
Record Dates: First submitted 2016-10-31; First posted 2016-11-01 (Estimated); Results first posted 2021-05-07 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Uveitis; Uveitis, Posterior; Uveitis, Anterior; Uveitis, Intermediate; Panuveitis
Keywords: Uveitis; UME; Posterior Uveitis; Anterior Uveitis; Intermediate Uveitis; Panuveitis; Non-infectious Uveitis; Triamcinolone; Choroid; Choroidal Injection; Suprachoroidal; Microneedle; Microinjection; Triamcinolone acetonide
MeSH Terms: conditions — Uveitis; Uveitis, Posterior; Uveitis, Anterior; Uveitis, Intermediate; Panuveitis | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 4 mg CLS-TA Suprachoriodal Injection: Those subjects randomized to the CLS-TA 4 mg arm in CLS1001-301 (NCT02595398) and who completed participation without receiving additional therapy. No study drug was administered during this study.
  Interventions: Drug: 4 mg CLS-TA Suprachoriodal Injection
- Sham procedure: Those subjects randomized to the sham procedure arm in CLS1001-301 (NCT02595398) and who completed participation without receiving additional therapy. No study drug was administered during this study.
  Interventions: Drug: Sham procedure

INTERVENTIONS:
Drug: 4 mg CLS-TA Suprachoriodal Injection — This drug was administered in the Parent study, CLS1001-301 (NCT02595398). No study treatments were administered during this observational extension study.
  Other Names: Triamcinolone Acetonide
  Groups: 4 mg CLS-TA Suprachoriodal Injection
Drug: Sham procedure — This drug was administered in the Parent study, CLS1001-301 (NCT02595398). No study treatments were administered during this observational extension study.
  Other Names: suprachoroidal sham
  Groups: Sham procedure

SUMMARY:
This study is a non-interventional, observational extension of the Parent study, CLS1001-301 (NCT02595398). The purpose of this study is to characterize the continued clinical benefit(s) regarding safety and efficacy of suprachoroidally administered CLS-TA, triamcinolone acetonide injectable suspension, for the treatment of macular edema associated with non-infectious uveitis.

DETAILED DESCRIPTION:
This is a non-interventional, observation extension study of up to 6 months for subjects completing the Parent study, CLS1001-301 (NCT02595398). The Parent study is a Phase 3, multicenter study to assess the safety and efficacy of 4 mg of CLS-TA administered via suprachoroidal injection compared to a sham procedure in the treatment of subjects with macular edema associated with non-infectious uveitis.

The design of the Extension study includes 4 clinic visits over a maximum of 24 weeks. Subject eligibility will be established at Visit 1 during the crossover day from the Parent study to the extension study (Day 0). Follow-up visits will be conducted every 6 weeks up to 24 weeks (Visit 4). At Visit 4, subjects will have a final evaluation conducted 24 weeks following study entry (48 weeks from Parent study randomization).

This study was initiated prior to the completion of the parent study, therefore treatment assignment was masked prior to study entry.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Parent study, CLS1001-301, through Visit 8/Month 6
* Willing and able to provide written informed consent prior to any study procedures; willing to comply with the instructions and attend all scheduled study visits

Exclusion Criteria:

* Received additional therapy for the treatment of uveitis or prohibited medication
* Require additional therapy for the treatment of uveitis or prohibited medication at the time of the Crossover visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include approximately 30 adult subjects that successfully complete the Parent study without requiring additional therapy to treat symptoms for uveitis as defined by the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ciulla, MD, Study Director — Clearside Biomedical, Inc.
Locations (16):
- United States (10):
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - Northern California Retina Vitreous Associates Medical Group, Inc., Mountain View, California
  - Retina Group of Florida, Fort Lauderdale, Florida
  - Marietta Eye Clinic, Marietta, Georgia
  - Valley Eye Physicians and Surgeons, PC, Ayer, Massachusetts
  - Bergstrom Eye Research, Fargo, North Dakota
  - Oregon Health & Science University Casey Eye Institute, Portland, Oregon
  - University of Pittsburgh Medical Center Eye Center, Pittsburgh, Pennsylvania
  - Texas Retina Associates, Dallas, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
- India (6):
  - Sri Sankaradeva Nethralaya, Guwahati, Assam
  - JSS Hospital, Mysore, Karnataka
  - Sankara Eye Hospital, Coimbatore, Tamil Nadu
  - King George's Medical University, Lucknow, Uttar Pradesh
  - Disha Eye Hospitals Pvt. Ltd., Kolkata
  - Dr Rajendra Prasad Centre for Ophthalmic Sciences, New Delhi

REFERENCES:
- [Derived] Yeh S, Ciulla T. Suprachoroidal triamcinolone acetonide injectable suspension for macular edema associated with noninfectious uveitis: an in-depth look at efficacy and safety. Am J Manag Care. 2023 Feb;29(2 Suppl):S19-S28. doi: 10.37765/ajmc.2023.89324. PMID 36787524

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled into the Parent study CLS1001-301 (NCT02595398), and who completed the Parent study without receiving additional therapy for uveitis were eligible for enrollment into this non-interventional observation extension study. The Parent study was still masked when subjects started enrolling into this extension study, therefore, treatment assignment was unknown at study entry and during the study.
Pre-assignment Details: Subjects enrolled into this non-interventional observational extension study successfully completed the Parent study CLS1001-301 (NCT02595398) without requiring additional therapy for uveitis. In the Parent study, subjects were randomized 3:2 to either 4 mg CLS-TA or a sham procedure in a masked fashion. Eligible and consenting subjects from selected sites were enrolled into the non-interventional extension study.
Groups:
- 4 mg CLS-TA Suprachoriodal Injection: Those subjects randomized to the CLS-TA 4 mg arm in CLS1001-301 (NCT02595398) and who completed participation in the Parent study without receiving additional therapy. No study drug was administered during this study.
  4 mg CLS-TA Suprachoriodal Injection: This drug was administered in the Parent study, CLS1001-301 (NCT02595398). No study treatments were administered during this observational extension study.
- Sham Procedure: Those subjects randomized to the sham procedure arm in CLS1001-301 (NCT02595398) and who completed participation in the Parent study without receiving additional therapy. No study drug was administered during this study.
  Sham procedure: This drug was administered in the Parent study, CLS1001-301 (NCT02595398). No study treatments were administered during this observational extension study.
Period: Overall Study
Arm/Group | 4 mg CLS-TA Suprachoriodal Injection | Sham Procedure
Started | 28 | 5
Completed | 14 | 2
Not Completed | 14 | 3
Not completed — Adverse Event | 3 | 0
Not completed — Prohibited therapy | 10 | 3
Not completed — Due to Posterior Capsular Opacity | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety population included all enrolled subjects who successfully completed the enrollment visit of the extension study.
Groups:
- Total: Total of all reporting groups
Arm/Group | 4 mg CLS-TA Suprachoriodal Injection | Sham Procedure | Total
Number analyzed (Participants) | 28 | 5 | 33
Age, Categorical [Count of Participants; unit: Participants] — Age of subjects in years relative to the date of the Screening visit from the Parent study CLS1001-301 (NCT02595398).
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 24 | 4 | 28
    >=65 years | 4 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of subjects in years relative to the date of the Screening visit from the Parent study CLS1001-301 (NCT02595398).
  years | 48.57 (15.039) | 51.20 (15.818) | 48.97 (14.934)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 1 | 15
  Male | 14 | 4 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 28 | 5 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 20 | 2 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 7 | 2 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 3 | 11
  India | 20 | 2 | 22
Type of Uveitis [Count of Participants; unit: Participants] — Location of inflammation in the study eye, including anterior (anterior chamber), intermediate (vitreous), posterior (retina or choroid) and panuveitis.
  Participants
    Anterior uveitis | 10 | 1 | 11
    Intermediate uveitis | 9 | 0 | 9
    Posterior uveitis | 11 | 1 | 12
    Panuveitis | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Time to Additional Therapy for Uveitis
Description: This time to event outcome was calculated as the number of days between the date of initiation of additional therapy for uveitis and the date of first treatment in the Parent study CLS1001-301 (NCT02595398).
Time Frame: 6 months following completion of the Parent study CLS1001-301 (NCT02595398), for a total of up to 1 year
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Groups:
- 4 mg CLS-TA Suprachoriodal Injection: Those subjects randomized to the CLS-TA 4 mg arm in CLS1001-301 (NCT02595398) and who completed participation i the Parent study without receiving additional therapy. No study drug was administered during this study.
  4 mg CLS-TA Suprachoriodal Injection: This drug was administered in the Parent study, CLS1001-301 (NCT02595398). No study treatments were administered during this observational extension study.
Arm/Group | 4 mg CLS-TA Suprachoriodal Injection | Sham Procedure
Number analyzed (Participants) | 28 | 5
days | 344.0 [282.0 to NA] — Not enough participants achieved response to calculate upper 95% CI | 332.0 [280.0 to NA] — Not enough participants achieved response to calculate upper 95% CI
Statistical Analysis 1: Comparison: 4 mg CLS-TA Suprachoriodal Injection vs Sham Procedure; The null hypothesis of no difference in the survival time distributions was tested; Test type: Superiority; p = 0.562, Log-rank chi-square test — The a priori threshold for statistical significance was 0.050. No adjustments made or required for multiplicity

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events and Serious Adverse Events
Description: Number of participants with treatment emergent adverse events and serious adverse events reported during the extension study.
Time Frame: 6 months following exit from Parent study
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | 4 mg CLS-TA Suprachoriodal Injection | Sham Procedure
Number analyzed (Participants) | 28 | 5
Participants
  Treatment-emergent adverse events | 16 | 3
  Serious adverse events | 1 | 0

3. Secondary Outcome: Mean Change From Baseline in Central Subfield Thickness
Description: Central subfield thickness (CST) is a diagnostic measurement used in identifying the presence of edema in the circular area 1 mm in diameter centered around the fovea. CST was measured using spectral domain optical coherence tomography (SD-OCT). A masked reading center graded the SD-OCT digital images. A negative change from baseline value represents a reduction in macular edema.
Time Frame: 6 months following exit from Parent study
Population: The Safety population included all enrolled subjects who successfully completed the enrollment visit of the extension study. Results include those subjects with gradable images at follow-up week 24. Values for missing data were not imputed.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | 4 mg CLS-TA Suprachoriodal Injection | Sham Procedure
Number analyzed (Participants) | 13 | 2
microns | -174.5 (145.70) | 19.5 (0.71)

4. Secondary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity
Description: Best corrected visual acuity (BCVA) refers to the measurement of the best possible vision that can be achieved following refraction or correction. BCVA was assessed following the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol and was measured in the number of letters read correctly on an ETDRS eye chart. An increase from the pre-treatment state in BCVA of 15 letters or more represents a clinically meaningful improvement.
Time Frame: 6 months following exit from Parent study
Population: The Safety population included all enrolled subjects who successfully completed the enrollment visit of the extension study. Results include those subjects with non-missing BCVA values at follow-up week 24. Values for missing data were not imputed.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | 4 mg CLS-TA Suprachoriodal Injection | Sham Procedure
Number analyzed (Participants) | 14 | 2
letters | 12.1 (13.00) | 14.0 (15.56)

ADVERSE EVENTS:
Time Frame: 6 months following completion of the Parent study CLS1001-301 (NCT02595398), for a total of up to 1 year.
Description: Treatment-emergent adverse events and SAEs initiating or worsening in severity relative to the date of enrollment into the extension study (day 0) were summarized.
Arm/Group | 4 mg CLS-TA Suprachoriodal Injection | Sham Procedure
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/5
Other Adverse Events (participants affected / at risk) | 16/28 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4 mg CLS-TA Suprachoriodal Injection (N=28) | Sham Procedure (N=5)
Oesophageal achalasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4 mg CLS-TA Suprachoriodal Injection (N=28) | Sham Procedure (N=5)
Infection parasitic (Infections and infestations) | 0 (0) | 1 (1)
Eosinophil count increased (Investigations) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 2 (2) | 0 (0) — #Study eye
Cataract cortical (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Cataract subcapsular (Eye disorders) | 5 (5) | 0 (0) — #Study eye
Macular fibrosis (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Macular oedema (Eye disorders) | 1 (1) | 1 (1) — #Study eye
Uveitis (Eye disorders) | 3 (3) | 1 (1) — #Study eye
Intraocular pressure increased (Investigations) | 3 (3) | 0 (0) — #Study eye
Cataract cortical (Eye disorders) | 0 (0) | 1 (1) — #Fellow eye
Eye pain (Eye disorders) | 2 (2) | 0 (0) — #Fellow eye
Uveitis (Eye disorders) | 2 (3) | 0 (0) — #Fellow eye

LIMITATIONS AND CAVEATS:
Subjects enrolled into the Parent study CLS1001-301 (NCT02595398), and who completed the Parent study without receiving additional therapy for uveitis were eligible for enrollment into this non-interventional observation extension study. The Parent study was still masked when subjects enrolled into this extension study, therefore, treatment assignment was unknown at study entry and remained masked until completion of the Parent study which occurred prior to the completion of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The institution and investigators participating in this trial shall have no right to publish or present the results of this study without the prior written consent of Clearside Biomedical.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-14): https://cdn.clinicaltrials.gov/large-docs/01/NCT02952001/Prot_SAP_000.pdf